CLINICAL TRIAL: NCT05253222
Title: Methodology and Clinical Value of Retrograde Imaging Technique in Intestinal Obstructive Diseases Mediated by Colonic Transendoscopic Enteral Tubing
Brief Title: Methodology and Clinical Value of RIT in Intestinal Obstructive Diseases Mediated by Colonic TET
Acronym: RIT;TET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other); Wuxi No. 2 People's Hospital (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TET2022N001
Record Dates: First submitted 2022-02-07; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Fecal Microbiota Transplantation; Bowel Obstruction
Keywords: Washed Microbiota Transplantation; Fecal Microbiota Transplantation; Transendoscopic enteral tubing
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- retrograde imaging by colonic TET (Experimental): Contrast fluid will be injected through colonic TET in participants with bowel obstruction. Image parameters detected by CT and X-ray fluoroscopy will be evaluated.
  Interventions: Diagnostic Test: retrograde image by colonic TET

INTERVENTIONS:
Diagnostic Test: retrograde image by colonic TET — Delivery of contrast fluid by colonic TET Each participant will receive one delivery of 200 ml contrast fluid by colonic TET to the distal portion of the lesion.
  One group will be taken CT investigation, another group will be taken X-ray fluoroscopy.
  Imaging parameters will be collected and evaluated.

SUMMARY:
The etiology of bowel obstruction is usually diagnosed by imaging techniques such as MSCTE,MRE, et al, which have some disadvantages. For example, in order to obtain better image quality, MSCTE（Multi-slices spiral computed tomography enterography） and MRE（ Magnetic resonance enterography）require patients to take a large amount of intestinal contrast solution orally, while for patients with intestinal obstruction, which may further aggravate the disease. Our study team had confirmed the mid-gut TET could serve as the delivery way of contrast solution for MRE bowel preparation with better accuracy of lesion detection and lower reduction of pain in CD（Crohn's Disease） patients. In this study, contrast solution will be delivered by colonic TET placed by lower GI-endoscopy, then we will evaluate the methodology and clinical value of this kind retrograde imaging technique in patients with intestinal obstructive diseases.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of intestinal obstruction such as abdominal pain, abdominal distension, nausea, vomiting, cessation of anal exhaust and defecation；
* Abdominal X-ray or plain CT showed signs of intestinal obstruction;
* Participants suspected with intestinal stricture according to the recent lower GI endoscopy；
* Voluntarily sign written informed consent.

Exclusion Criteria:

* Signs of peritonitis, perforation or massive hemorrhage of digestive tract;
* Accompanied with severe heart, brain, lung and kidney dysfunction, unable to take lower GI endoscopy;
* Allergic to laxatives or iodine contrast agents;
* Pregnant women;
* Confirmed or suspected claustrophobia;
* Inability to understand or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic self-confidence score | immediately after CT/X-ray fluoroscopy detection，no more than 24hours.
  Image parameters of the lesion( i e. Location，Nature, Severity, Appearance, Fistula) will be recorded by the reader.
  The diagnostic self-confidence for each image parameter will be determined using a continuous five-grade scoring system from 1 to 5(1 = worst, 2=worsen, 3=normal, 4= better,5 = best).
  For example:
  The doctor's diagnostic self-confidence for Location is worsen ,then the diagnostic self-confidence score will be recorded as 2。
Evaluation of comprehensive diagnostic efficiency | immediately after CT/X-ray fluoroscopy detection，no more than 24hours.
  comprehensive diagnostic efficiency=(Location+Nature+Appearance+Fistula+Proximal lesion filled by contrast fluid）. Each positive parameter will be recorded as mark 1, negative mark 0. Each participant will get up to 5 score.
  For example:
  for some one participant ,if the doctor could determine the location and nature of the lesion, however,appearance, fistula and proximal lesion filled by contrast fluid could not be determined, then ,the score of comprehensive diagnostic efficiency equals 2.

SECONDARY OUTCOMES:
Adverse reaction | during the process, and no more than 24hours after CT/X-ray fluoroscopy detection
  Adverse reaction( abdominal pain, abdominal distention, nausea, vomiting) will be recorded and graded by score 1 to 5 according to the severity of each symptom.
Tolerance | during the process, and no more than 24hours after CT/X-ray fluoroscopy detection
  Tolerance will be evaluated by questionnaire investigation。1--Severely intolerable；2--Moderately intolerable；3--Slightly intolerable；4--Tolerable。

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD, PhD, Study Chair — Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rami Reddy SR, Cappell MS. A Systematic Review of the Clinical Presentation, Diagnosis, and Treatment of Small Bowel Obstruction. Curr Gastroenterol Rep. 2017 Jun;19(6):28. doi: 10.1007/s11894-017-0566-9. PMID 28439845
- [Background] Catena F, De Simone B, Coccolini F, Di Saverio S, Sartelli M, Ansaloni L. Bowel obstruction: a narrative review for all physicians. World J Emerg Surg. 2019 Apr 29;14:20. doi: 10.1186/s13017-019-0240-7. eCollection 2019. PMID 31168315
- [Background] Sheedy SP, Kolbe AB, Fletcher JG, Fidler JL. Computed Tomography Enterography. Radiol Clin North Am. 2018 Sep;56(5):649-670. doi: 10.1016/j.rcl.2018.04.002. Epub 2018 Jul 11. PMID 30119766
- [Background] Masselli G, Gualdi G. CT and MR enterography in evaluating small bowel diseases: when to use which modality? Abdom Imaging. 2013 Apr;38(2):249-59. doi: 10.1007/s00261-012-9961-8. PMID 23011551
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Background] Dai M, Zhang T, Li Q, Cui B, Xiang L, Ding X, Rong R, Bai J, Zhu J, Zhang F. The bowel preparation for magnetic resonance enterography in patients with Crohn's disease: study protocol for a randomized controlled trial. Trials. 2019 Jan 3;20(1):1. doi: 10.1186/s13063-018-3101-x. PMID 30606236